CLINICAL TRIAL: NCT00786526
Title: Ventilator-Induced Diaphragmatic Dysfunction (VIDD) in Critically Ill Patients
Brief Title: Diaphragmatic Function in Ventilated Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF7854
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Critically Ill
Keywords: Mechanical ventilation; Ventilator induced diaphragmatic dysfunction; Weaning; Neuromuscular diseases- Respiratory function tests; Intubated patients in intensive care unit
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Animal studies showed that controlled mechanical ventilation (CMV) can induce dysfunction of the diaphragm, resulting in an early-onset and progressive decrease in diaphragmatic force-generating capacity, called ventilator-induced diaphragmatic dysfunction (VIDD).

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation (tracheally intubated or tracheotomized) less than 48h.·
* Duration of mechanical ventilation for at least 72h.·
* Subject itself or its next of kin has given written informed consent

Exclusion Criteria:

* Patient is less than 18 years or more than 85 years of age·
* The attending physician refuses to allow enrollment·
* The patient refuses informed consent
* Next of kin is unavailable or refuses informed consent·
* Pregnant or breast-feeding female.
* A pregnancy test will be performed in all female patients less than 60 years of age.·
* Any contraindication to use cervical magnetic stimulation (mechanical cardiac assist device …).·
* Presence or suspicion of prior diaphragm injury or chronic disease·
* Presence or suspicion of a central nervous system (CNS) disorder, including (but not limited to): CNS infarction, bleeding, tumor, or infection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated patients in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2008-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Respiratory function parameters | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas SIMILOWSKI, MD, PhD, Study Chair — Groupe Hospitalier La Pitié-Salpêtrière-Paris
Locations (2):
- France (2):
  - Department of Anesthesia and Critical Care (DAR B), Saint-Eloi University Hospital of Montpellier, Montpellier
  - Service de Pneumologie et Réanimation, Groupe Hospitalier La Pitié-Salpêtrière-Paris, Paris

REFERENCES:
- [Derived] Demoule A, Molinari N, Jung B, Prodanovic H, Chanques G, Matecki S, Mayaux J, Similowski T, Jaber S. Patterns of diaphragm function in critically ill patients receiving prolonged mechanical ventilation: a prospective longitudinal study. Ann Intensive Care. 2016 Dec;6(1):75. doi: 10.1186/s13613-016-0179-8. Epub 2016 Aug 5. PMID 27492005
- [Derived] Demoule A, Jung B, Prodanovic H, Molinari N, Chanques G, Coirault C, Matecki S, Duguet A, Similowski T, Jaber S. Diaphragm dysfunction on admission to the intensive care unit. Prevalence, risk factors, and prognostic impact-a prospective study. Am J Respir Crit Care Med. 2013 Jul 15;188(2):213-9. doi: 10.1164/rccm.201209-1668OC. PMID 23641946